CLINICAL TRIAL: NCT05755841
Title: Inpatient Versus Outpatient Management of Preterm Prelabour Rupture of Membrane. A Prospective Cohort Study
Brief Title: Outpatient Management of Preterm Prelabor Rupture of Membranes
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer in Obstetrics and Gynecology, Ain Shams Maternity Hospital
Other Study IDs: 9
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Management of Preterm Prelabor Rupture of Membranes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Outpatient management of preterm prelabor rupture of membranes
  Interventions: Other: Outpatient management of preterm prelabor rupture of membranes
- 2: Inpatient management of preterm prelabor rupture of membranes
  Interventions: Other: Inpatient management of preterm prelabor rupture of membranes

INTERVENTIONS:
Other: Outpatient management of preterm prelabor rupture of membranes — Patients who will be managed as outpatients will be discharged after 48 hours of hospitalization with the following management:
  * Twice weekly fetal cardiotocography.
  * Complete blood count once a week.
  * A weekly clinical and ultrasound examination.
  Groups: 1
Other: Inpatient management of preterm prelabor rupture of membranes — In the Inpatient Care Policy group, the same protocol as outpatient group will be applied, but the patient will not be discharged until delivery.
  Groups: 2

SUMMARY:
Home-care management is possible if patients are clinically stable forty-eight hours after Preterm Prelabour Rupture of the membrane with no clinical or biological signs suggestive of intrauterine infection. Several retrospective studies have highlighted the safety of such outpatient management for women with nonthreatening Preterm Prelabour Rupture of the membrane. This prospective cohort study will compare inpatient versus outpatient management of preterm Prelabour rupture of membrane regarding latency, intra-amniotic infection, birth weight, and neonatal complications at 28 to 34 weeks of gestation after 48 hours of admission to Ain-Shams University Maternity Hospital.

DETAILED DESCRIPTION:
The fetal membranes are made of two histological layers, the amnion in contact with the amniotic fluid, and the chorion in contact with the maternal decidua. They engrave the fetus during pregnancy and serve as a barrier between the maternal and fetal compartments, supplying both physicochemical and biochemical defense against external shocks and rising vaginal flora bacteria.

Membrane rupture is a biochemical phenomenon that happens towards the conclusion of birth. The programmed weakening of the Para cervical region, marked by collagen remodeling and apoptosis coupled with uterine contractions that produce stretching and shearing forces, contributes to the breakup of the membranes.

The rupture that happens before initiating contractions in 10% of pregnancies is called "Prelabour membrane rupture" (PROM). About 3% of women undergo Prelabour Rupture of the membrane before 37 weeks of birth, which is considered preterm pre-labor membrane breakup (PPROM). This condition is responsible for one-third of preterm births and raises perinatal morbidity and mortality primarily due to the risk of intrauterine infection, which may lead to early neonatal infection, necrotizing enterocolitis, and uterine fetal death

In spite of major progress in antenatal management over the past three decades, Prelabour membrane rupture and prenatal birth are still common. About 50 percent of women with Preterm Prelabour Rupture of the membrane (<37 WG) bear children within 24-48 hours after rupture and 70 percent to 90 percent within 7 days. Patients with Preterm Prelabour Rupture of the membrane need clinical treatment in a hospital that has the required services for premature babies. When the point of fetal viability is met, Preterm Prelabour Rupture of the membrane is initially hospital-based and consists of antibiotic prophylaxis and corticosteroids for fetal lung maturation. The key surveillance priorities are the diagnosis and treatment of maternal and fetal complications, in particular intrauterine infections. Home-care treatment is possible if patients are clinically stable 48 hours post Prelabour Rupture of the membrane with no clinical or biological symptoms of intrauterine infection. The protection of such outpatient management for women with non-threatening Preterm Prelabour Rupture of the membrane has been illustrated in many retrospective studies.

Home-care inclusion requirements are based on gestational age, lack of chorioamnionitis, physiological reliability at least 72 hours after Preterm Prelabour Rupture of the membrane (up to 7 days depending on the study), cervical dilation, and patient at home. The time between membrane breakup and labor initiation, referred to as latency, is stated to be correlated with neonatal morbidity and mortality. While certain factors, such as gestational age at Preterm Prelabour Rupture of the membrane, cervical dilation, parity, twin pregnancy, and chorioamnionitis, have been reported to affect latency in the literature, the time between rupture and delivery remains difficult to predict. Awareness of short-term predictive variables could optimize the length of hospital stay and help forecast the likelihood of adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 28-34 weeks as calculated from the Last Menstrual period, Ultrasound examination in early 2nd trimester at 14 weeks, or first trimetric ultrasound.
2. Confirmed preterm Prelabour rupture of membranes using a Sterile Cusco speculum examination, definitive history of gush of watery discharge or ultrasound measurement of the deepest vertical pocket <2cm.

Exclusion Criteria:

1. Mutiple pregnancy
2. Cases with congenital fetal malformations conditioning prognosis
3. Preterm prelabor rupture of membranes associated with preeclampsia, Diabetes mellitus, Systemic lupus erythematosus, long term steroid therapy, Renal/hepatic impairment
4. Preterm Prelabour Rupture of membrane-associated with antepartum hemorrhage or asymptomatic Placenta Previa
5. Past history of classic Cesarean section

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women admitted to Ain Shams University Maternity Hospital due to preterm prelabor rupture of membranes
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Latency period | From the time of membrane rupture till the time of delivery
  the interval between rupture of the membranes and the onset of labor.

SECONDARY OUTCOMES:
Intraamniotic infection | From the time of membrane rupture till the time of delivery
  ▪ Intra-amniotic infection, will be diagnosed clinically :
  * Maternal fever >38°c.
  * Purulent cervical discharge.
  * Fetal tachycardia>160 beats/min.
Birth weight | First 24 hours after delivery
  Neonatal birth weight

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

REFERENCES:
- [Background] Richardson L, Kim S, Menon R, Han A. Organ-On-Chip Technology: The Future of Feto-Maternal Interface Research? Front Physiol. 2020 Jun 30;11:715. doi: 10.3389/fphys.2020.00715. eCollection 2020. PMID 32695021
- [Background] Kumar D, Moore RM, Mercer BM, Mansour JM, Redline RW, Moore JJ. The physiology of fetal membrane weakening and rupture: Insights gained from the determination of physical properties revisited. Placenta. 2016 Jun;42:59-73. doi: 10.1016/j.placenta.2016.03.015. Epub 2016 Apr 1. PMID 27238715
- [Background] Mercer, B.M. (2012), I240 MANAGEMENT OF PTL/PPROM. International Journal of Gynecology & Obstetrics, 119: S221-S221
- [Background] Souza RT, Cecatti JG. A Comprehensive Integrative Review of the Factors Associated with Spontaneous Preterm Birth, Its Prevention and Prediction, Including Metabolomic Markers. Rev Bras Ginecol Obstet. 2020 Jan;42(1):51-60. doi: 10.1055/s-0040-1701462. Epub 2020 Feb 27. PMID 32107766
- [Background] Hume, Robert. (2014). The Value of Money in Eighteenth-Century England: Incomes, Prices, Buying Power-and Some Problems in Cultural Economics. Huntington Library Quarterly. 77. 373-416.
- [Background] Schmitz T, Sentilhes L, Lorthe E, Gallot D, Madar H, Doret-Dion M, Beucher G, Charlier C, Cazanave C, Delorme P, Garabedian C, Azria E, Tessier V, Senat MV, Kayem G. Preterm premature rupture of the membranes: Guidelines for clinical practice from the French College of Gynaecologists and Obstetricians (CNGOF). Eur J Obstet Gynecol Reprod Biol. 2019 May;236:1-6. doi: 10.1016/j.ejogrb.2019.02.021. Epub 2019 Mar 2. PMID 30870741
- [Background] Guckert M, Clouqueur E, Drumez E, Petit C, Houfflin-Debarge V, Subtil D, Garabedian C. Is homecare management associated with longer latency in preterm premature rupture of membranes? Arch Gynecol Obstet. 2020 Jan;301(1):61-67. doi: 10.1007/s00404-019-05363-x. Epub 2019 Nov 23. PMID 31760462
- [Background] Ministry of Health. 2021. Induction of Labour in Aotearoa New Zealand: A clinical practice guideline 2019. Wellington: Ministry of Health
- [Background] Kibel M, Asztalos E, Barrett J, Dunn MS, Tward C, Pittini A, Melamed N. Outcomes of Pregnancies Complicated by Preterm Premature Rupture of Membranes Between 20 and 24 Weeks of Gestation. Obstet Gynecol. 2016 Aug;128(2):313-320. doi: 10.1097/AOG.0000000000001530. PMID 27400016
- [Background] Bouchghoul H, Kayem G, Schmitz T, Benachi A, Sentilhes L, Dussaux C, Senat MV. Outpatient versus inpatient care for preterm premature rupture of membranes before 34 weeks of gestation. Sci Rep. 2019 Mar 12;9(1):4280. doi: 10.1038/s41598-019-40585-8. PMID 30862787
- [Background] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050